CLINICAL TRIAL: NCT05159323
Title: Quantitative Parameters of Diffusion Spectrum Imaging: Correlation With Histopathologic Characteristics in Patients With Breast Cancer
Brief Title: Quantitative Assessment of Diffusion Spectrum Imaging in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiang Zhang (Other)
Responsible Party: Sponsor-Investigator, Xiang Zhang, Department of Radiology, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SYSEC-KY-KS-2021-182
Record Dates: First submitted 2021-11-21; First posted 2021-12-16 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Breast Carcinoma; Magnetic Resonance Imaging; Diffusion Spectrum Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diffusion Spectrum Imaging (Experimental): All participants accept diffusion spectrum imaging, the quantitative parameters of the diffusion spectrum imaging are obtained. The quantitative parameters are compared in different subgroups based on the pathologic examination results.
  Interventions: Diagnostic Test: Diffusion Spectrum Imaging

INTERVENTIONS:
Diagnostic Test: Diffusion Spectrum Imaging — A novel diffusion-based magnetic resonance imaging method

SUMMARY:
This project intends to prospectively collect patients with suspected breast malignant tumors by ultrasound or mammography. After routine MRI scanning, all patients underwent diffusion spectrum imaging (DSI) sequence scanning. The inclusion criteria were as follows: (1) breast cancer was confirmed by surgery or biopsy. (2) pathologically diagnosis of estrogen receptor (ER), progesterone receptor (PR), human epidermal growth factor 2 (HER-2), Ki-67, and lymphatic vessel invasion (LVI) status in breast cancer. (3) routine MRI and DSI scans were performed within one week before the pathologic examination. The exclusion criteria were as follows: (1) patients who had received treatment before DSI scanning; (2) patients who underwent breast tumor biopsy within two weeks before DSI image acquisition; (3) pathology results of breast masses were other diseases besides breast cancer. (4) post-processing of DSI data cannot be performed due to poor image quality, such as motion artifacts.

Breast MRI data were collected on a 3T MR scanner (Magnetom skyra, Siemens Healthcare, Erlangen, Germany). All participants used standardized breast MRI scanning schemes, including T2 weighted imaging (T2WI), T1 weighted imaging (T1WI), diffusion-weighted imaging (DWI), DSI, and contrast dynamic enhancement (DCE). A total of 22 GSI quantitative parameters were derived from NeudiLab software that is based on the open-source platform DIPY (diffusion imaging in Python, http://nipy.org/dipy). The correlation between DSI quantitative parameters and pathological indexes (i.e., ER, PR, HER-2, Ki-67, and LVI) was evaluated by Spearman correlation analysis. The independent predictors of GSI quantitative parameters for different pathologic characteristics discrimination in breast cancer were determined by the logistic regression analysis. The predictive performance of DSI quantitative parameters for difference pathologic classifications was assessed by the receiver operating characteristic (ROC) curves and their respective area under the curves (AUCs).

ELIGIBILITY:
Inclusion Criteria:

1. Breast cancer was confirmed by surgery or biopsy.
2. Pathologically diagnosis of estrogen receptor (ER), progesterone receptor (PR), human epidermal growth factor 2 (HER-2), Ki-67, and lymphatic vessel invasion (LVI) status in breast cancer.
3. Routine MRI and DSI scans were performed within one week before the pathologic examination.

Exclusion Criteria:

1. Patients who had received treatment before DSI scanning.
2. Patients who underwent breast tumor biopsy within two weeks before DSI image acquisition.
3. Pathology results of breast masses were other diseases besides breast cancer.
4. Post-processing of DSI data cannot be performed due to poor image quality, such as motion artifacts.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-08-19 (Estimated); Study Completion 2022-08-19 (Estimated)

PRIMARY OUTCOMES:
Pathologic characteristic | Up to 2 months
  Estrogen receptor (ER) status of breast cancer

SECONDARY OUTCOMES:
Pathologic characteristic | Up to 2 months
  Progesterone receptor (PR) status of breast cancer

OTHER OUTCOMES:
Pathologic characteristic | Up to 2 months
  Human epidermal growth factor 2 (HER-2) status of breast cancer
Pathologic characteristic | Up to 2 months
  Ki-67 status of breast cancer
Pathologic characteristic | Up to 2 months
  Lymphatic vessel invasion (LVI) status of breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Zhang, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Radiology, Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Qiu Y, Jiang W, Yang Z, Wang M, Li Q, Liu Y, Yan X, Yang G, Shen J. Mean Apparent Propagator MRI: Quantitative Assessment of Tumor-Stroma Ratio in Invasive Ductal Breast Carcinoma. Radiol Imaging Cancer. 2024 Jul;6(4):e230165. doi: 10.1148/rycan.230165. PMID 38874529